CLINICAL TRIAL: NCT01067443
Title: A Phase II Randomized, Parallel Arm, Open-labeled Clinical Trial to Assess the Safety and Efficacy of the Combination of Sodium Stibogluconate Plus Single Dose AmBisome®, Miltefosine Plus Single Dose AmBisome® and Miltefosine Alone for the Treatment of Primary Visceral Leishmaniasis in Eastern Africa
Brief Title: Clinical Trial to Assess the Safety and Efficacy of Sodium Stibogluconate (SSG) and AmBisome® Combination, Miltefosine and AmBisome® and Miltefosine Alone for the Treatment Visceral Leishmaniasis in Eastern Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Gilead Sciences (Industry); Paladin Labs Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEAP 0208
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Primary Visceral Leishmaniasis
Keywords: Phase II; Randomised clinical trial; Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B; Antimony Sodium Gluconate; miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amb+SSG (Experimental): AmBisome® one dose of 10mg/kg body weight (IV) on day 1 followed by 10 days of SSG at 20mg/kg body weight (IV/IM) from days 2-11
  Interventions: Drug: Liposomal amphotericin B (AmBisome®) and sodium stibogluconate
- Amb+Milt (Experimental): AmBisome® one dose of 10mg/kg body weight (IV) on day 1 followed by 10 days Miltefosine at 2.5mg/kg body weight (oral) from days 2-11
  Interventions: Drug: Liposomal amphotericin B + miltefosine
- Milt (Experimental): Monotherapy course of Miltefosine at 2.5mg/kg body weight (oral) from days 1-28
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Liposomal amphotericin B (AmBisome®) and sodium stibogluconate — AmBisome® one dose of 10mg/kg body weight (IV) on day 1 followed by 10 days of SSG at 20mg/kg body weight (IV/IM) from days 2-11
  Arms: Amb+SSG
Drug: Liposomal amphotericin B + miltefosine — AmBisome® one dose of 10mg/kg body weight (IV) on day 1 followed by 10 days Miltefosine at 2.5mg/kg body weight (oral) from days 2-11
  Arms: Amb+Milt
Drug: Miltefosine — Monotherapy course of Miltefosine at 2.5mg/kg body weight (oral) from days 1-28
  Arms: Milt

SUMMARY:
This study is to assess if shorter combinations of SSG plus single dose AmBisome®, Miltefosine plus single dose AmBisome® and Miltefosine alone are effective in treating visceral leishmaniasis in Eastern Africa.

DETAILED DESCRIPTION:
The current study intends to look at potential feasible short course combination therapies as well as evaluate (and possibly register) miltefosine in its conventional dose against VL in Sudan and Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical signs and symptoms of VL and diagnosis confirmed by visualization of parasites in tissue samples (lymph node, bone marrow or spleen where relevant) on microscopy.
* Patients aged between 7 (to allow for blood sampling) and 60 years (inclusive) who are able to comply with the protocol.
* Patients for whom written informed consent has been signed by the patients themselves (if aged 18 years and over) or by parents(s) or legal guardian for patients under 18 years of age.
* HIV negative status

Exclusion Criteria:

* Patients who have received any anti-leishmanial drugs in the last 6 months/ relapse cases.
* Patients with a negative lymph node/bone marrow (or spleen) smears.
* Patients with severe protein and or caloric malnutrition (Kwashiorkor or marasmus ; Adults: BMI </= 15, Children W/H<70, presence of oedema)
* Patients with previous history of hypersensitivity reaction to SSG or Amphotericin B.
* Patients suffering from a concomitant severe infection such as TB or any other serious underlying disease (cardiac, renal, hepatic) which would preclude evaluation of the patient's response to study medication.
* Patients suffering from other conditions associated with splenomegaly such as schistosomiasis.
* Patients with previous history of cardiac arrhythmia or an abnormal ECG
* Patients who are female of child bearing age (all females who have achieved menarche) / pregnant or lactating.
* Patients with haemoglobin < 5gm/dl.
* Patients with WBC < 1 x 10³/mm³.
* Patients with platelets < 40,000/mm³.
* Patients with abnormal liver function (ALT and AST) tests of more than three times the normal range.
* Patients with serum creatinine outside the normal range for age and gender.
* Major surgical intervention within 2 weeks prior to enrolment.

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Initial cure: proportion cured at Day 28 | Day 28

SECONDARY OUTCOMES:
Final cure: proportion cured at day 210 | 6 months post treatment
Adverse events and serious adverse events occurring in the three study arms | up to day 60

CONTACTS AND LOCATIONS:
Overall Officials: Monique Wasunna, MD, Principal Investigator — Kenya Medical Research Institute
Locations (3):
- Kimalel Health Centre, Kimalel, Kenya
- Sudan (2):
  - Kassab Hospital, Kassāb, Al Qaḑārif
  - El Hassan Centre for Tropical Medicine, Doka, Gedarif

REFERENCES:
- [Derived] Wasunna M, Njenga S, Balasegaram M, Alexander N, Omollo R, Edwards T, Dorlo TP, Musa B, Ali MH, Elamin MY, Kirigi G, Juma R, Kip AE, Schoone GJ, Hailu A, Olobo J, Ellis S, Kimutai R, Wells S, Khalil EA, Strub Wourgaft N, Alves F, Musa A. Efficacy and Safety of AmBisome in Combination with Sodium Stibogluconate or Miltefosine and Miltefosine Monotherapy for African Visceral Leishmaniasis: Phase II Randomized Trial. PLoS Negl Trop Dis. 2016 Sep 14;10(9):e0004880. doi: 10.1371/journal.pntd.0004880. eCollection 2016 Sep. PMID 27627654
- [Derived] Allison A, Edwards T, Omollo R, Alves F, Magirr D, E Alexander ND. Generalizing boundaries for triangular designs, and efficacy estimation at extended follow-ups. Trials. 2015 Nov 16;16:522. doi: 10.1186/s13063-015-1018-1. PMID 26573827
- [Derived] Omollo R, Alexander N, Edwards T, Khalil EA, Younis BM, Abuzaid AA, Wasunna M, Njoroge N, Kinoti D, Kirigi G, Dorlo TP, Ellis S, Balasegaram M, Musa AM. Safety and efficacy of miltefosine alone and in combination with sodium stibogluconate and liposomal amphotericin B for the treatment of primary visceral leishmaniasis in East Africa: study protocol for a randomized controlled trial. Trials. 2011 Jun 30;12:166. doi: 10.1186/1745-6215-12-166. PMID 21718522
- Available data/document: Study Protocol — http://journals.plos.org/plosntds/article/file?type=supplementary&id=info:doi/10.1371/journal.pntd.0004880.s002 — Final Study Protocol